CLINICAL TRIAL: NCT01001845
Title: Comparative Effects of Milk Thistle Extract With Vitamin-E on Oxidative Stress Biomarkers in Hemodialysis Patients
Brief Title: Comparative Effects of Milk Thistle Extract With Vitamin-E in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Dr. Jamshid Roozbeh, Nephrology and Urology Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 53001
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2010-09

CONDITIONS: Hemodialysis; End Stage Renal Disease
Keywords: hemodialysis; oxidative stress; plasma malondialdehyde; Glutathion peroxidase
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — milk-thistle extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lifestyle counseling (No Intervention)
- vit E (Active Comparator): 200mg 2 times per day for 3 weeks
  Interventions: Drug: vit E
- Milk Thistle extract (Experimental): 1 tablet (equivalent to 140 mg silymarin) 3 times a day for 3 weeks
  Interventions: Drug: Milk Thistle extract
- vit E + Milk Thistle Extract (Experimental): 200mg vit E twice a day + 1 tablet of Milk Thistle extract 3 times a day for 3 weeks
  Interventions: Drug: vit E + Milk Thistle extract

INTERVENTIONS:
Drug: Milk Thistle extract — 1 tablet equivalent to 140 mg of silymarin, 3 times daily for 3 weeks
  Arms: Milk Thistle extract
Drug: vit E — 200 mg twice daily for 3 weeks
  Arms: vit E
Drug: vit E + Milk Thistle extract — 200 mg vit E twice daily + 1 tablet of Milk Thistle 3 times daily for 3 weeks
  Arms: vit E + Milk Thistle Extract

SUMMARY:
For end-stage renal disease (ESRD) patients, cardiovascular disease remains the single most common cause of excess morbidity and mortality. Among the examined nontraditional risk factors, an increase in oxidative stress as well as inflammation are postulated to contribute to excessive cardiovascular risk in this population.

Flavonoids are naturally occurring substances that possess various pharmacological actions and therapeutic applications. Some due to their phenolic structures have antioxidant effect and inhibit free radical-mediated processes, as well as anti-inflammatory effects. Silymarin,a mixture of three isomeric flavonolignans, is isolated from milk thistle (Silybum marianum) seeds, and is proven to have anti-oxidant, anti-inflammatory, cell regenerating, and antifibrotic action.

In this study, the effect of silymarin on oxidative stress and inflammation (2 major risk factors for cardiovascular morbidity and mortality in hemodialysis patients)is evaluated, and compared to vit E, a well known antioxidant.

ELIGIBILITY:
Inclusion Criteria:

* All hemodialysis patients age 18-60
* On hemodialysis for over 3 months, 3 times a week, and for 4 hours each time
* Signed informed consent

Exclusion Criteria:

* Heart Failure NYHA Class III or IV
* Recent MI (within 1 year)
* Use of anti-oxidant supplements: N-acetyl-cystein, Omega 3, Vit C, Vit E, green tea, soy extracts, pomegranate extract, grape extract..
* Hepatitis B or C
* Active Infection
* Psychiatric illness
* Active malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
RBC Glutathion Peroxidase level | 3 weeks

SECONDARY OUTCOMES:
Plasma malondialdehyde | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ghazal Vessal, PharmD, PhD, Study Director — Shiraz University of Medical Sciences, Faculty of Pharmacy; Bahram Shahriari, MD, Principal Investigator — Shiraz University of Medical Sciences; Jamshid Roozbeh, MD, Study Chair — Nephrology Urology Research Center, Shiraz University of Medical Sciences; masoumeh Akmali, PhD, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Nemazi Hospital, Shiraz, Fars, Iran